CLINICAL TRIAL: NCT00002473
Title: A Prospective Randomized Phase III Study Comparing Radical Surgery to Elective Kidney Sparing Surgery for Low Stage Renal Cell Carcinoma
Brief Title: Kidney-Sparing Surgery Compared With Kidney Removal in Treating Patients With Kidney Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Eastern Cooperative Oncology Group (Network); American College of Surgeons (Other); SWOG Cancer Research Network (Network); NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: EORTC-30904; EORTC-30904; ACOSOG-30904; CAN-NCIC-RE1; E-30904; SWOG-EORTC-30904
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2013-06

CONDITIONS: Kidney Cancer
Keywords: stage I renal cell cancer; stage II renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell

INTERVENTIONS:
Procedure: conventional surgery

SUMMARY:
RATIONALE: Kidney-sparing surgery is a less invasive type of surgery for kidney cancer, and may have fewer side effects and improve recovery. It is unknown whether kidney-sparing surgery is more effective than kidney removal in treating kidney cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of surgery to completely remove the kidney with kidney-sparing surgery in treating patients with resectable kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare time to recurrence and survival of patients with single, low stage, nonmetastatic, well localized, and well delineated renal cell cancer treated with partial vs radical resection.
* Establish the side effects of kidney-sparing tumor resection in terms of morbidity and mortality in these patients.
* Study the relationship between tumor size, histologic grade, histologic type, and the extent of local control following partial resection.
* Determine which prognostic factors are important in selecting candidates for conservative surgery.

OUTLINE: This is a randomized, multicenter study.

Patients are randomized to undergo radical nephrectomy and limited lymphadenectomy (arm I) or conservative surgery (arm II).

Patients are followed every 3 months for 1 year, every 4 months for 2 years, every 6 months for 2 years, then annually thereafter.

PROJECTED ACCRUAL: A total of 1300 patients will be accrued for this study over 8 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Single renal T1-2 tumor suspicious for adenocarcinoma that meets the following requirements:

  * Solitary tumor on CT scan
  * Maximum diameter 5 cm
  * Located such that negative resection margins are assured
  * N0, M0, i.e., no nodal involvement or distant metastases

    * No invasion of renal pelvis, calices, or perirenal fat as determined by CT scan or intravenous urography
  * Normal contralateral kidney present
* No von Hippel-Lindau disease

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* WHO 0-2

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* No second malignancy except adequately treated nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-03; Primary Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hein van Poppel, MD, PhD, Study Chair — University Hospital, Gasthuisberg; Thomas Keane, MD, Study Chair — Emory University; Leonard G. Gomella, MD, Study Chair — Sidney Kimmel Cancer Center at Thomas Jefferson University; Eila C. Skinner, MD, Study Chair — University of Southern California; Laurence H. Klotz, MD, Study Chair — Toronto Sunnybrook Regional Cancer Centre
Locations (2):
- Canada (2):
  - Sunnybrook and Women's College Health Sciences Centre, North York, Ontario
  - McGill University, Montreal, Quebec

REFERENCES:
- [Result] Van Poppel H, Da Pozzo L, Albrecht W, Matveev V, Bono A, Borkowski A, Colombel M, Klotz L, Skinner E, Keane T, Marreaud S, Collette S, Sylvester R. A prospective, randomised EORTC intergroup phase 3 study comparing the oncologic outcome of elective nephron-sparing surgery and radical nephrectomy for low-stage renal cell carcinoma. Eur Urol. 2011 Apr;59(4):543-52. doi: 10.1016/j.eururo.2010.12.013. Epub 2010 Dec 22. PMID 21186077
- [Result] Van Poppel H, Da Pozzo L, Albrecht W, Matveev V, Bono A, Borkowski A, Marechal JM, Klotz L, Skinner E, Keane T, Claessens I, Sylvester R; European Organization for Research and Treatment of Cancer (EORTC); National Cancer Institute of Canada Clinical Trials Group (NCIC CTG); Southwest Oncology Group (SWOG); Eastern Cooperative Oncology Group (ECOG). A prospective randomized EORTC intergroup phase 3 study comparing the complications of elective nephron-sparing surgery and radical nephrectomy for low-stage renal cell carcinoma. Eur Urol. 2007 Jun;51(6):1606-15. doi: 10.1016/j.eururo.2006.11.013. Epub 2006 Nov 15. PMID 17140723
- [Derived] Scosyrev E, Messing EM, Sylvester R, Van Poppel H. Exploratory Subgroup Analyses of Renal Function and Overall Survival in European Organization for Research and Treatment of Cancer randomized trial of Nephron-sparing Surgery Versus Radical Nephrectomy. Eur Urol Focus. 2017 Dec;3(6):599-605. doi: 10.1016/j.euf.2017.02.015. Epub 2017 Apr 4. PMID 28753863
- [Derived] Scosyrev E, Messing EM, Sylvester R, Campbell S, Van Poppel H. Renal function after nephron-sparing surgery versus radical nephrectomy: results from EORTC randomized trial 30904. Eur Urol. 2014 Feb;65(2):372-7. doi: 10.1016/j.eururo.2013.06.044. Epub 2013 Jul 2. PMID 23850254